CLINICAL TRIAL: NCT05133440
Title: SAXON-PC: A Phase II Randomized Trial of Stereotactic Body Radiation Therapy (SBRT) And Radium (Ra-223) Dichloride for Oligorecurrent, Non-castrate Resistant Prostate Cancer
Brief Title: A Study of Stereotactic Body Radiation Therapy and Radium (Ra-223) Dichloride in Prostate Cancer That Has Spread to the Bones
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-213
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; SBRT; Non-castrate Resistant Prostate Cancer; Oligorecurrent Prostate Cancer; SAXON-PC; 21-213; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride; Radium-223; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Participants will receive two cycles of Radium (Ra-223) dichloride at 55 kBq/kg or 0.00149 mCi/kg or 1.49 uCi/kg every 4 weeks followed 2-3 weeks later by SBRT at a dose of 9 Gy per fraction for 3 fractions (total dose of 27 Gy) to all sites of radiographically apparent metastatic disease. SBRT to the target index lesion(s) should be completed within 30 days after simulation after completion of the 2nd infusion of Radium (Ra-223) dichloride. Specific dose constraints, dosing schedules, and management of SBRT to multiple sites will be at the discretion of the treating Radiation oncologist. The goal is to complete simulation and SBRT within 30 days. Only active or progressive disease is to be treated at the discretion of the treating investigator.
  Interventions: Drug: Radium dichloride
- Control Arm: (Active Comparator): Participants will receive SBRT at a dose of 9 Gy per fraction for 3 fractions (total dose of 27 Gy) to all sites of radiographically apparent metastatic disease. SBRT fractions can be administered every day or every other day per institutional practice. SBRT should begin within 30 days (+/- 7 days) of randomization. Only active or progressive disease is to be treated at the discretion of the treating investigator.
  Interventions: Drug: Radium dichloride; Diagnostic Test: PET Scan

INTERVENTIONS:
Drug: Radium dichloride — Two cycles of Radium (Ra-223) dichloride at 55 kBq/kg or 0.00149 mCi/kg or 1.49 uCi/kg every 4 weeks followed 2-3 weeks later by SBRT at a dose of 9 Gy per fraction for 3 fractions (total dose of 27 Gy) to all sites of radiographically apparent metastatic disease. SBRT fractions can be administered every day or every other day per institutional practice. An additional 4 cycles of Radium (Ra-223) dichloride at 55 kBq/kg or 0.00149 mCi/kg or 1.49 uCi/kg every 4 weeks will then be administered, resuming 2-3 weeks after completion of the final fraction of SBRT.
  Other Names: Ra-223
Diagnostic Test: PET Scan — For both arms, the NaF PET will be used to identify discrete osseous lesions which will become index lesions for the study. The simulation scan (either baseline or after 2 cycles of Ra-223) will be used to generate a suitable SBRT radiation plan, per standard practice. If the index lesions are no longer visible after two cycles of Ra-223, we still intend to consolidate the area with radiation. If the lesions are initially radio-occult on the CT and only visible on the NaF PET, we will fuse the pre-treatment NaF PET/CT to the simulation CT after 2 cycles of Ra-223 to delineate the SBRT treatment volumes.
  Other Names: NaF PET
  Arms: Control Arm:

SUMMARY:
Participants will either receive treatment with standard SBRT and the study drug Radium (Ra-223) dichloride, or standard SBRT alone.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma
* ≥ 18 years old
* Primary prostate tumor must have been treated with prior prostatectomy or definitive radiotherapy
* Men with prior salvage radiotherapy to the prostate bed and/or locoregional lymph nodes are eligible assuming normalization of testosterone
* Negative multi-parametric MRI and/or negative biopsy of the prostate (or prostate bed) within 60 days of enrollment
* Pre-enrollment imaging (any bone imaging modality per institutional standard of care) demonstrates oligometastatic disease with 1-3 discrete metastatic lesions of the bone performed within 60 days of study enrollment; screening PSMA PET confirming 1-3 sites of oligometastatic disease performed within 60 days of enrollment.
* All bony oligometastatic sites must be deemed appropriate to receive 3 fraction SBRT to a dose of 9 Gy x 3 at best judgment of treating radiation oncologist
* Prostate specific antigen (PSA) ≥ 0.5 ng/mL but ≤ 50 ng/mL
* Patients may have had prior androgen deprivation therapy (ADT) but must have normal testosterone levels (>100 ng/dL) at time of enrollment; patients with baseline low testosterone but no ADT exposure are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Subjects who have not had surgical removal of their prostate and have a partner of child bearing potential must agree to use condoms beginning at the signing of the consent until at least 6 months after the last dose of study drug. Because of the potential side effect on spermatogenesis associated with radiation, female partners of childbearing potential must agree to use a highly effective contraceptive method during and for 6 months after completing treatment. Examples of highly effective contraception options for women include implantable uterine devices (hormonal or non-hormonal), oral, patch and parenteral contraceptives (when taken as prescribed).
* Adequate hematological, liver and renal function

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelet count ≥ 100 x 10^9/L
  * Hemoglobin ≥ 10.0 g/dL
  * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Creatinine ≤ 1.5 x ULN with normal creatinine clearance
  * Albumin > 25 g/L
* Patient willing and able to comply with the protocol, including follow-up visits and examination

Exclusion Criteria:

* Pathological findings consistent with small cell and/or neuroendocrine carcinoma of the prostate or any other histology
* Any metastatic site >5 cm in maximum diameter
* Patients with documented castration resistant prostate cancer (CRPC)
* Patients with any form of conventional, metabolic or molecular imaging (including PET imaging with PSMA, fluciclovine and/or FDG tracers) within 60 days of enrollment that demonstrate more than 3 discrete metastatic lesions
* Patients with evidence of nonpelvic lymph nodal or any visceral metastases
* Patients with evidence of progressing locoregional lymph nodes (prior lymphadenectomy or definitive/salvage RT to the pelvic lymph nodes is acceptable assuming no evidence of progression)
* Patients with documented or suspected impending significant spinal cord compression defined as epidural spinal cord compression (ESCC) grade 2 or higher using the Bilsky scale
* Patients with parenchymal brain metastases
* Patient received any other investigational therapeutic agents or other anticancer therapeutics within 4 weeks prior to randomization
* Major surgery within 30 days prior to start of study drug
* Any prior systemic therapy with radionuclide agents (e.g., strontium-89, samarium-153, rhenium-186, rhenium-188 or Radium (Ra-223) dichloride) for the treatment of bony metastases
* Fecal incontinence
* History of another malignancy within the previous 3 years except for the following:

adequately treated basal cell or squamous cell skin cancer

* Any other serious illness or medical condition, such as but not limited to:

  * Any infection greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v 5.0 Grade 2
  * New York Heart Association (NYHA) Class III or IV heart failure
  * Crohn's disease or ulcerative colitis
  * Bone marrow dysplasia or myelodysplastic syndrome

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2027-11-12 (Estimated); Study Completion 2027-11-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  The primary outcome is to compare rates of composite PFS between the two treatment arms using bone scan imaging. A patient will be considered to have disease progression if any of the following events occur from the time of protocol randomization to date of last follow-up: a) PSA biochemical progression OR b) Radiographical progression OR c) clinical progression OR d) start of ADT OR e) death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Imber, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - University of Colorado (Data Collection Only), Aurora, Colorado
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org